CLINICAL TRIAL: NCT02826694
Title: North Carolina Newborn Exome Sequencing for Universal Screening
Acronym: NC_NEXUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Human Genome Research Institute (NHGRI) (NIH); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-2409; 5U19HD077632 (NIH)
Record Dates: First submitted 2016-06-21; First posted 2016-07-11 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2019-03

CONDITIONS: Metabolism, Inborn Errors; Hearing Loss; Hereditary Disease
MeSH Terms: conditions — Metabolism, Inborn Errors; Hearing Loss; Genetic Diseases, Inborn | interventions — Exome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Well infant, whole exome sequencing (Other): Healthy infants and their parents enrolled in the study prenatally will participate. After the infant is born saliva sample will be collected for DNA extraction and whole exome sequencing will be done.
  Interventions: Genetic: Well infant, whole exome sequencing
- Diagnosed, whole exome sequencing (Other): Infants and children with diagnosed conditions whose parents enroll in the study and consent to having their child sequenced will have saliva samples obtained and whole exome sequencing will be done on extracted DNA.
  Interventions: Genetic: Diagnosed, whole exome sequencing

INTERVENTIONS:
Genetic: Well infant, whole exome sequencing — Whole exome sequencing will be performed in children with diagnosed conditions. Investigators will analyze results that are associated with their condition.
  Arms: Well infant, whole exome sequencing
Genetic: Diagnosed, whole exome sequencing — In addition to returning results of conditions associated with a child's phenotype, investigators will also analyze genes that are associated with conditions that have childhood onset and are medically actionable.
  Arms: Diagnosed, whole exome sequencing

SUMMARY:
The NC NEXUS research study is exploring the utility of next generation sequencing in newborn screening and parental decision making. The National Institutes of Health (NICHD and NHGRI) are co-funding this study under a single U-19.

DETAILED DESCRIPTION:
The investigators will enroll and perform whole exome sequencing on two cohorts of patients. One cohort will consist of two hundred newborns with no known conditions whose parents will be recruited during the mother's pregnancy. The second cohort will include two hundred infants and children up to the age of five years with diagnosed conditions including conditions detected through standard newborn screening such as phenylketonuria and other inborn errors of metabolism, hearing loss and other rare conditions that may fit criteria for newborn screening in the future.

Parents will be introduced to the study by their clinician or a study recruiter. Those who agree to enroll in Phase I will review an online decision guide and be offered a study visit conducted by a genetic counselor to obtain informed consent for genomic sequencing of their child. Parents consenting to have their child's genome sequenced will be seen after the child's birth or at a convenient pre-arranged time and duplicate saliva samples will be collected from the children and one sample will be sent to the BioSpecimen Processing (BSP) Facility and to Dr. Jonathan Berg's laboratory for sequencing and the other sent to the Molecular Genetics Laboratory (MGL) for DNA extraction and storage until needed for clinical confirmation. Results will be returned for diagnostic (in the Diagnosed cohort) and medically actionable disorders of childhood (both cohorts). Two-thirds of parents who consent to sequencing will be randomly assigned to be eligible to request additional findings and use a supplement of the online decision aid. All results will be reported to parents by trained genetic professionals (genetic counselors and clinical geneticists)

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated pregnancy and healthy newborn

Exclusion Criteria:

* Abnormalities such as major malformation or chromosomal disorder detected prenatally or significant complications during pregnancy or at the time of delivery.

Ages: 1 Hour to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2016-06; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Berg, MD, PhD, Principal Investigator — University of North Carolina School of Medicine Department of Genetics; Cynthia M Powell, MD, Principal Investigator — University of North Carolina School of Medicine Department of Pediatrics
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Sequencing data will be shared via the Newborn Screening Translational Research Network.

REFERENCES:
- [Derived] Milko LV, Rini C, Lewis MA, Butterfield RM, Lin FC, Paquin RS, Powell BC, Roche MI, Souris KJ, Bailey DB Jr, Berg JS, Powell CM. Evaluating parents' decisions about next-generation sequencing for their child in the NC NEXUS (North Carolina Newborn Exome Sequencing for Universal Screening) study: a randomized controlled trial protocol. Trials. 2018 Jun 28;19(1):344. doi: 10.1186/s13063-018-2686-4. PMID 29950170

RESULTS

PARTICIPANT FLOW:
Groups:
- Well Infant, Whole Exome Sequencing: Healthy infants and their parents enrolled in the study prenatally will participate. After the infant is born saliva sample will be collected for DNA extraction and whole exome sequencing will be done. Investigators will analyze results associated with childhood onset, medically actionable conditions.
- Diagnosed, Whole Exome Sequencing: Infants and children with diagnosed conditions whose parents enroll in the study and consent to having their child sequenced will have saliva samples obtained and whole exome sequencing will be done on extracted DNA. In addition to returning results of conditions associated with the child's phenotype, investigators will also analyze genes that are associated with conditions that have childhood onset and are medically actionable.
Period: Overall Study
Arm/Group | Well Infant, Whole Exome Sequencing | Diagnosed, Whole Exome Sequencing
Started | 61 | 45
Decision Group | 41 | 30
Control Group | 20 | 15
Completed | 61 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy newborns and children up to age 5 with a diagnosed condition
Groups:
- Well Infant, Whole Exome Sequencing: Healthy infants and their parents enrolled in the study prenatally will participate. After the infant is born saliva sample will be collected for DNA extraction and whole exome sequencing will be done. Investigators will analyze genes that are associated with conditions that have childhood onset and are medically actionable.
- Total: Total of all reporting groups
Arm/Group | Well Infant, Whole Exome Sequencing | Diagnosed, Whole Exome Sequencing | Total
Number analyzed (Participants) | 61 | 45 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 61 | 45 | 106
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 32 | 17 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 51 | 42 | 93
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 44 | 37 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 45 | 106

OUTCOME MEASURES:

1. Primary Outcome: Parental Choices Following Decision Aid
Description: Analysis of parents' decisions after they complete an on-line decision aid to see if they wish to participate in the study. Options will be yes, no, or undecided.
Time Frame: average of 3-6 months
Population: Those parents initially approached received an email link to the 1st Decision Aid. However, they were not considered enrolled unless they came for an in-person consent visit and elected to have their child's genome sequenced.
Measure: Count of Participants; unit: Participants
Arm/Group | Well Infant, Whole Exome Sequencing | Diagnosed, Whole Exome Sequencing
Number analyzed (Participants) | 145 | 59
Participants
  Said yes or undecided after decision aid | 120 | 57
  Did not want child sequenced | 25 | 2

2. Primary Outcome: Number of Participants Identified With Genetic Conditions Through Whole Exome Sequencing
Description: Investigators analyzed next generation sequencing (NGS) results in the diagnosed cohort to determine the ability of whole exome sequencing to detect pathogenic variants in genes related to phenotype determined by standard newborn screening (NBS). The category of genes analyzed is termed the Next Generation Sequencing/Newborn Screening (NGS/NBS) category. Healthy newborns with no known genetic conditions also had the NGS/NBS category of genes analyzed.
Time Frame: approximately 3-6 months after DNA sample obtained
Population: By definition, there were no well infants in the "Diagnosed, whole exome sequencing" Arm category.
Measure: Count of Participants; unit: Participants
Arm/Group | Well Infant, Whole Exome Sequencing | Diagnosed, Whole Exome Sequencing
Number analyzed (Participants) | 61 | 45
Participants
  All participants: Well infant | 61 | 0
  All participants: Hearing Loss | 0 | 28
  All participants: Metabolic Disorder | 0 | 17
  Positive NGS/NBS result: number analyzed (Participants) | 1 | 20
  Positive NGS/NBS result: Well infant | 1 | 0
  Positive NGS/NBS result: Hearing Loss | 0 | 5
  Positive NGS/NBS result: Metabolic Disorder | 0 | 15
  Negative NGS/NBS results: number analyzed (Participants) | 60 | 25
  Negative NGS/NBS results: Well infant | 60 | 0
  Negative NGS/NBS results: Hearing Loss | 0 | 23
  Negative NGS/NBS results: Metabolic Disorder | 0 | 2

3. Secondary Outcome: Parental Reaction Scores
Description: Test-related distress is assessed with an adapted version of the Multidimensional Impact of Cancer Risk Assessment (MICRA). It asks participants to report how often in the past week they have experienced worries and distress related to their child's genomic sequencing procedure and test results, and the social and familial consequences of sequencing and the test results. Possible responses are provided on the following scale: 0=Never, 1=Rarely, 3=Sometimes, and 5=Often. Because it refers to respondents' experience of their child's sequencing and the test results they received, it is administered only in assessments that occurred after sequencing at Time 3 (2 weeks after results visit and Time 4 (3 months after results visit). Comparisons are made between couples who could chose to receive additional information about their child's genome and a control group who were not eligible to receive additional information.
Time Frame: Time 3 - 2 weeks after results visit and Time 4 - 3 months after results visit
Population: Total number completing T3 and T4 MICRA scales
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Decision Arm: 2/3 of families from both groups of the study (Well Infant and Diagnosed) were randomized into the Decision Arm that could learn additional information from results of their child's genome sequencing (childhood onset non-medically actionable conditions, adult onset actionable conditions, or carrier status). "Families" include single mothers or couples. Numbers indicate total number who completed the time 3 and time 4 distress measure.
- Control Arm: 1/3 of families from both groups of the study (Well Infant and Diagnosed) were randomized into the Control Arm and did not receive the option of additional information from their child's genome sequencing. "Families" include single mothers or couples. Numbers indicate total number who completed the time 3 and time 4 distress measure.
Arm/Group | Decision Arm | Control Arm
Number analyzed (Participants) | 126 | 54
score on a scale
  T3 | 2.3 (2.4) | 1.7 (1.5)
  T4 | 2.5 (2.5) | 1.5 (0.4)
Statistical Analysis 1: Comparison: Decision Arm vs Control Arm; T3; Test type: Other; p = 0.168, linear mixed effect model
Statistical Analysis 2: Comparison: Decision Arm vs Control Arm; T4; Test type: Other; p = 0.026, linear mixed effect model

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning at Baseline and continued through Time 4 (3 months after results visit).
Arm/Group | Well Infant, Whole Exome Sequencing | Diagnosed, Whole Exome Sequencing
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/45
Other Adverse Events (participants affected / at risk) | 0/61 | 2/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Well Infant, Whole Exome Sequencing (N=61) | Diagnosed, Whole Exome Sequencing (N=45)
Sample mixup (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT02826694/Prot_SAP_000.pdf